CLINICAL TRIAL: NCT04936568
Title: Implementation of a Standardized Palliative Care Referral System (PCRS) for Cancer Patients With Advanced Disease: Impact on Patient and Caregiver Satisfaction With Care and Use of Health Care Resources.
Brief Title: Palliative Care Referral System (PCRS) for Cancer Patients With Advanced Disease
Acronym: PCRSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Augusto Caraceni, director of Palliative Care Unit, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201/19
Record Dates: First submitted 2021-06-08; First posted 2021-06-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Cancer
Keywords: early palliative care; referral

STUDY DESIGN:
Intervention Model Description: A quasi-experimental, longitudinal, pretest-posttest study will be carried out. Two different cohorts of 150 advanced cancer patients each will be enrolled before (pretest) and after (posttest) the introduction of the PCRS in outpatient clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): standard oncology care
- intervention (Experimental): standardized referral to outpatient palliative care by oncologists
  Interventions: Other: Palliative Care Referral System - PCRS

INTERVENTIONS:
Other: Palliative Care Referral System - PCRS — Implementation of a system to help oncologists to identify criteria for referring patients to specialized outpatient palliative care (Palliative Care Referral System - PCRS)
  Arms: intervention

SUMMARY:
Early palliative care (EPC) in the clinical pathway of advanced cancer patients improves symptom control, quality of life and has a positive impact on overall quality of care. EPC contributes to realistic and attainable goals of treatment, facilitating patient choices, favouring adequate communication with patients and families and assessing patient values and preferences with regard to advance care planning. EPC is likely to promote a more appropriate use of health care resources and less aggressive cancer treatment in the last weeks of life. At present standardised criteria for appropriate referral for EPC in oncology outpatients setting are lacking. Therefore the aim of this project is to identify referral criteria and procedures to implement appropriate EPC for advanced patients (the Palliative Care Referral System) and test them in a pre-post experimental design evaluating their impact on quality of care and on the use of healthcare resources. A quasi-experimental, longitudinal, pretest-posttest study will be carried out. Two different cohorts of 150 advanced cancer patients each will be enrolled before (pretest) and after (posttest) the introduction of the PCRS in outpatient clinics of a Comprehensive Cancer Centre. Eligible patients will undergo patient-reported outcome measure (PROMs) evaluation at baseline and then monthly for at least 6 months from enrollment or till death. Use health care resources and quality of care indicators will be collected monthly by a dedicated research nurse.

DETAILED DESCRIPTION:
As above.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years;
* recent diagnosis of inoperable locally advanced and/or metastatic cancer not eligible to anticancer treatment with curative intent;

Exclusion Criteria:

* cognitive impairment that would prevent self-assessments
* current palliative care treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
patient reported experience | through study completion, up to 6 months
  patient satisfaction with care, measured with the FAMCARE-P13

SECONDARY OUTCOMES:
Health related quality of life | through study completion, up to 6 months
  European Organisation for Research and Treatment of Cancer - Quality of Life -Palliative Care questionnaire (Eortc QLQC15-PAL)
caregiver experience of care | through study completion, up to 6 months
  Family Care Satisfaction scale (FAMCARE)
Activation of a Palliative Care service | through study completion, up to 6 months
  Number of regular outpatient Palliative Care visits
Multidisciplinary team visits | through study completion, up to 6 months
  Number of multidisciplinary team visits (Oncology and Palliative Care)
Hospitalization | through study completion, up to 6 months
  Number of hospitalizations
Emergency department accesses | through study completion, up to 6 months
  Number of accesses in Emergency departement

CONTACTS AND LOCATIONS:
Overall Officials: Augusto T Caraceni, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
not planned

REFERENCES:
- [Derived] Brunelli C, Zecca E, Pigni A, Bracchi P, Caputo M, Lo Dico S, Fusetti V, Tallarita A, Bergamini C, Brambilla M, Raimondi A, Niger M, Provenzano S, Sepe P, Alfieri S, Tine G, De Braud F, Caraceni AT. Outpatient palliative care referral system (PCRS) for patients with advanced cancer: an impact evaluation protocol. BMJ Open. 2022 Oct 28;12(10):e059410. doi: 10.1136/bmjopen-2021-059410. PMID 36307164